CLINICAL TRIAL: NCT04888962
Title: Quantitative Sensory Psychophysical Correlates of Pain in Pregnant Women With OUD
Acronym: Q-PRONTO
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Grace Lim, MD, MS, Associate Professor, University of Pittsburgh
Other Study IDs: STUDY20060069
Record Dates: First submitted 2021-05-11; First posted 2021-05-17 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-10

CONDITIONS: Opioid-use Disorder; Pregnancy Related
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prospective cohort group: This cohort will include pregnant patients with a history of opiate use disorder (OUD) who will be followed from the third trimester of pregnancy until 24 hours postpartum.
  Interventions: Other: OUD
- Control group: This cohort will include pregnant patients without a history of opiate use disorder (OUD) who will be followed from the third trimester of pregnancy until 24 hours postpartum.

INTERVENTIONS:
Other: OUD — History of opioid use disorder.
  Groups: Prospective cohort group

SUMMARY:
This is a prospective observational case-control study comparing quantitative sensory testing data preformed during the third trimester of pregnancy and within 24 hours postpartum in women on medication-assisted treatment for opioid use disorder (OUD) to a gestational age-controlled cohort of women who do not have OUD.

The primary goal is to measure elements of quantitative sensory testing including temperature pain threshold, temperature pain tolerance, and thermal and mechanical temporal summation for patients with opioid use disorder on medication-assisted treatment (MAT), and compare these results to gestational age matched controlled pregnant patients not on MAT.

DETAILED DESCRIPTION:
The objective of this study is to measure elements of quantitative sensory testing including temperature pain threshold, temperature pain tolerance, and thermal and mechanical temporal summation for patients with opioid use disorder on medication-assisted treatment (MAT), and compare these results to gestational age matched controlled pregnant patients not on MAT.

The hypothesis is that women requiring maintenance opioids during pregnancy will have a significant difference in pain sensitivity in the third trimester and immediately postpartum as compared to women who did not require maintenance opioids during pregnancy.

ELIGIBILITY:
Inclusion Criteria:

Subjects that will be included in the prospective cohort group:

* individuals at least 18 years of age
* at least 28 weeks gestation (third trimester)
* on medication-assisted treatment for opioid use disorder, including methadone or suboxone.

Patients who will be included in the control group:

* individuals at least 18 years of age
* at least 28 weeks gestation (third trimester)
* have not been on been on opioids in the past 12 months.

Exclusion Criteria:

* Those who are unable to participate in informed consent discussions,
* Unable to give informed consent for any reason,
* Not fluent in English (surveys are validated in English language)
* Unable to participate fully in all study procedures for any reason including sensory deficits, scar tissue, or infection at any QST sites.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will enroll pregnant adults with opiate use disorder (on medication assisted therapy) who are currently in their third trimester.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2021-06-14 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
QST Pain threshold | Completed at a time point antepartum/ before delivery
  Quantitative sensory testing is a pain sensitivity test in which the patient will tell the investigator the moment they first feel pain
QST Pain Tolerance | Completed at a time point antepartum/ before delivery
  Quantitative sensory testing is a pain sensitivity test in which the patient will tell the investigator the moment the sensation becomes uncomfortable.
QST Pain Threshold | Completed within 24 hours postpartum/ after delivery
  Quantitative sensory testing is a pain sensitivity test in which the patient will tell the investigator the moment they first feel pain
QST Pain Tolerance | Completed within 24 hours postpartum/ after delivery
  Quantitative sensory testing is a pain sensitivity test in which the patient will tell the investigator the moment the sensation becomes uncomfortable.

CONTACTS AND LOCATIONS:
Overall Officials: Grace Lim, MD, MS, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No